CLINICAL TRIAL: NCT01417780
Title: Evaluation of Safety, Pharmacokinetics and Immunomodulatory Effects of AB103, a CD28 Co-stimulatory Receptor Antagonist, in Patients Diagnosed With Necrotizing Soft Tissue Infections
Brief Title: Evaluation of Safety, PK and Immunomodulatory Effects of AB103 in Necrotizing Soft Tissue Infections Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atox Bio Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATB-201
Record Dates: First submitted 2011-08-11; First posted 2011-08-16 (Estimated); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Necrotizing Soft Tissue Infections
MeSH Terms: interventions — AB103

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AB103 0.25 mg/kg (Active Comparator)
  Interventions: Drug: AB103
- AB103 0.5 mg/kg (Active Comparator)
  Interventions: Drug: AB103
- Placebo (Placebo Comparator): Normal saline (0.9% sodium chloride)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AB103 — AB103 0.25 mg/kg or 0.5 mg/kg administered as a single IV infusion
  Other Names: p2TA
  Arms: AB103 0.25 mg/kg; AB103 0.5 mg/kg
Drug: Placebo — Normal saline (0.9% sodium chloride) administered as a single IV infusion
  Arms: Placebo

SUMMARY:
A study to evaluate the safety and pharmacokinetics profile of different doses of AB103 administered to patients diagnosed with Necrotizing Soft Tissue Infections that are scheduled for an urgent surgical intervention as part of their standard of care.

DETAILED DESCRIPTION:
A study to evaluate the safety and pharmacokinetics profile of different doses of AB103 administered to patients diagnosed with Necrotizing Soft Tissue Infections that are scheduled for an urgent surgical intervention as part of their standard of care. The primary study hypothesis is that AB-103 can be administered safely to the patients presenting with Necrotizing Soft Tissue Infections.

Secondary endpoints are efficacy by exploratory descriptive analyses of specific efficacy endpoints from three outcome domains to demonstrate treatment benefit of AB103 in comparison to placebo in patients with Necrotizing Soft Tissue Infections. The efficacy domains are:

1. Clinical status domain
2. Pharmacoeconomics domain
3. Systemic and local inflammatory biomarker domain

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of NSTI due to bacterial infection (Necrotizing Fasciitis, Group A streptococcal infection or non group A streptococcal infection, Fournier's gangrene, Bacterial synergistic gangrene, Synergistic Necrotizing Cellulitis, Clostridial gas gangrene/ myonecrosis) that may be supported by specific signs and symptoms, e.g. tense edema outside area of compromised skin, pain disproportionate to appearance, skin discoloration, ecchymosis, blisters/bullae, necrosis, tense edema, crepitus and/or subcutaneous gas AND a decision for urgent surgical exploration and debridement;
* Patient who did not receive the study drug prior to the surgery need to have a definite diagnosis of NSTI confirmed surgically (e.g. presence of necrotic tissue, thrombosed vessels in the subcutaneous tissue, lack of bleeding and "dishwater" (cloudy, thin, gray) fluid) in order to get the drug during or after operation;
* IV drug administration within 6 hours from the clinical diagnosis and from the documented decision to have an urgent surgical exploration and debridement;
* Signed and dated ICF as defined by the IRB and, if applicable, California Bill of Rights. By signing the ICF, the patient agrees to release any medical records pursuant to current Health Insurance Portability and Accountability Act (HIPAA) Guidelines. If patient is unable to comprehend or sign the ICF, patient's legally acceptable representative may sign the ICF;

Exclusion Criteria

* Age < 18 years;
* Weight > 150 Kg / 330 pounds;
* Pregnant or lactating women; Female of childbearing potential, the patient must have a negative beta subunit hCG pregnancy test immediately prior to study entry (performed by urine or blood test, whichever is faster);
* Patient who has been operated at least once for the current NSTI infection and had a curative deep tissue debridement (diagnostic surgery is allowed to enter into the study);
* Known HIV infection with CD4 count < 200 cells/mm3 or < 14% of all lymphocytes;
* Diabetic patients with below ankle infection;
* Patients with overt peripheral vascular disease in the involved area - condition associated with ischemic ulcers and /or symptoms of inadequate vascular supply (e.g. intermittent claudication) where limb amputation is considered likely within 7 days;
* Current status of: a. Mean arterial pressure < 50 mmHg and/or systolic blood pressure < 70 mmHg despite treatment with vasopressors and/or IV fluids or b. a patient with respiratory failure such that an SaO2 of 80% cannot be achieved or c. a patient with refractory coagulopathy (INR > 3) or d. thrombocytopenia (platelet count < 20,000) that does not partially correct with administration of appropriate factors, or e. likely severe neurological impairment secondary to cardiac arrest.
* Patients with cardiac arrest requiring cardiopulmonary resuscitation within the past 30 days;
* Patient is not expected to survive 30 days because of underlying medical condition, such as poorly controlled neoplasm (e.g. Stage III or IV cancer);
* Any concurrent medical condition, which in the opinion of the investigator, may compromise their safety or the objectives of the study or the patient will not benefit from treatment, (e.g. end stage organ disease {CHF {NYHA class III-IV}, COPD {stage III-IV}, Liver dysfunction {Childs-Pugh class C}, Renal dysfunction {Dialysis}), immunosuppression, receiving or about to receive chemotherapy or known severe neutropenia < 1,000 cells/mm3;
* Patients with Necrotizing Soft Tissue Infection post intra-abdominal operation;
* Patient with burn wounds;
* Patient or patient's family are not committed to aggressive management of the patient's condition, or the combination of necrotizing skin infection and underlying illness makes it unlikely that life support will be maintained;
* Previous enrolment in an previous clinical trial involving investigational drug or a medical device within 30 days before provision of written informed consent for the study or within five half lives of the investigational drug, whichever is longer;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Southern California Los Angeles, Los Angeles, California
  - San Francisco General Hospital, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bulger EM, Maier RV, Sperry J, Joshi M, Henry S, Moore FA, Moldawer LL, Demetriades D, Talving P, Schreiber M, Ham B, Cohen M, Opal S, Segalovich I, Maislin G, Kaempfer R, Shirvan A. A Novel Drug for Treatment of Necrotizing Soft-Tissue Infections: A Randomized Clinical Trial. JAMA Surg. 2014 Jun;149(6):528-36. doi: 10.1001/jamasurg.2013.4841. PMID 24740134
- [Result] Bulger EM, Maislin G, Dankner W, May A, Edgar R, Shirvan A. Critical Care Medicine, January 2018,46(1):327. Abstract 682: Early Plasma Cytokine Levels Correlate With Outcome in Necrotizing Soft Tissue Infections. https://journals.lww.com/ccmjournal/Citation/2018/01001/682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by qualified investigators under the sponsorship of Atox Bio Ltd. at 7 trauma centers, of which 6 enrolled patients from December 2011 through August 2012.
Pre-assignment Details: Of 43 randomized patients who received AB103 or placebo (intent-to-treat [ITT] population; safety analyses), 3 patients were excluded to form the modified intent-to-treat (mITT) population before unblinding due to protocol violations. Therefore, a total of 40 patients were included in the mITT efficacy analyses. With respect to any variable, the number of patients analyzed is the number of patients with non-missing data within the respective population.
Groups:
- AB103 0.25 mg/kg: AB103 0.25 mg/kg administered as a single IV infusion
- AB103 0.5 mg/kg: AB103 0.5 mg/kg administered as a single IV infusion
Period: Overall Study
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Started (ITT Population) | 15 | 17 | 11
Completed (ITT Population) | 14 | 14 | 9
Not Completed | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Data are from the modified intent-to-treat (mITT) population. The mITT population consisted of all randomized patients who received the proper study drug (AB103 or placebo) and dose, had a definitive surgical diagnosis of NSTI, and did not have a CD4 count <200 cells/mm3.
Groups:
- Total: Total of all reporting groups
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.6) | 50.1 (15.2) | 52.5 (20.4) | 50.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 14
  Male | 11 | 9 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 13 | 14 | 9 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 14 | 14 | 7 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
NSTI Diagnosis [Count of Participants; unit: Participants]
  Fournier Gangrene | 5 | 6 | 2 | 13
  Other NSTI | 10 | 9 | 8 | 27
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.0 (6.5) | 31.7 (9.7) | 29.9 (9.3) | 31.5 (8.2)
Acute Physiology And Chronic Health Evaluation II (APACHE II) Score [Mean (Standard Deviation); unit: units on a scale] — APACHE II is a severity of illness classification system. It is determined within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements (physiologic variables, age, chronic health status).
  Higher scores correspond to more severe disease and a greater risk of death.
  units on a scale | 7.5 (5.0) | 8.3 (4.5) | 9.6 (4.7) | 8.3 (4.7)
Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — SOFA total scores range from 0 to 24, with higher scores reflecting a worse clinical status or outcome. A SOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
  units on a scale | 2.87 (2.70) | 3.47 (2.53) | 3.10 (1.97) | 3.15 (2.42)
Cardiovascular Organ Failure [Count of Participants; unit: Participants] | 1 | 4 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With One or More Adverse Events (AEs) During the Treatment Period
Description: An AE is any untoward medical occurrence in a subject administered study drug and that does not necessarily have a causal relationship with the study drug. An AE could therefore be any unfavorable and unintended sign (including abnormal laboratory findings), symptom, or disease temporally associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: 7 days
Population: The safety analysis population consisted of all randomized patients who received study drug (N=43). The number of patients analyzed is the number of patients with non-missing data in this population.
Measure: Count of Participants; unit: Participants
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 17 | 11
Participants | 14 | 16 | 9

2. Primary Outcome: Number of Subjects With One or More Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is an AE occurring during any study phase and at any dose of the study drug (AB103 or placebo) that fulfills one or more of the following criteria:
  * Results in death
  * Is life-threatening (i.e., the subject was, in the opinion of the Investigator, at immediate risk of death from the event as it occurred)
  * Requires or prolongs hospitalization
  * Results in persistent or significant disability or incapacity (i.e., the event causes a substantial disruption of a person's ability to conduct normal life functions)
  * Is a congenital anomaly or birth defect, or
  * Is an important and significant medical event.
Time Frame: 28 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 17 | 11
Participants | 8 | 5 | 4

3. Primary Outcome: Alanine Aminotransferase (ALT)
Description: Screening ALT results, Day 7 ALT results, and change in ALT from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 12 | 15 | 10
units/L
  Screening | 55.9 (99.8) | 28.1 (17.3) | 46.8 (57.2)
  Day 7: number analyzed (Participants) | 10 | 12 | 9
  Day 7 | 27.9 (18.8) | 27.3 (26.3) | 26.0 (13.2)
  Change from Screening to Day 7: number analyzed (Participants) | 10 | 12 | 9
  Change from Screening to Day 7 | -23.2 (95.1) | -0.8 (31.2) | -19.8 (60.5)

4. Primary Outcome: Aspartate Aminotransferase (AST)
Description: Screening AST results, Day 7 AST results, and change in AST from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 17 | 11
units/L
  Screening | 35.8 (30.6) | 37.4 (28.3) | 32.0 (19.2)
  Day 7: number analyzed (Participants) | 10 | 12 | 9
  Day 7 | 30.6 (17.1) | 24.3 (10.1) | 27.4 (9.7)
  Change from Screening to Day 7: number analyzed (Participants) | 10 | 12 | 9
  Change from Screening to Day 7 | -1.2 (30.7) | -9.3 (21.7) | 0.1 (9.6)

5. Primary Outcome: Alkaline Phosphatase (ALP)
Description: Screening ALP results, Day 7 ALP results, and change in ALP from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/L
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 17 | 11
units/L
  Screening | 97.5 (53.5) | 104.3 (47.7) | 108.3 (44.2)
  Day 7: number analyzed (Participants) | 10 | 12 | 8
  Day 7 | 93.1 (45.2) | 84.8 (33.9) | 100.6 (65.9)
  Change from Screening to Day 7: number analyzed (Participants) | 10 | 12 | 8
  Change from Screening to Day 7 | 5.2 (40.1) | -10.6 (62.3) | -11.4 (34.6)

6. Primary Outcome: Total Bilirubin (Tbili)
Description: Screening Tbili results, Day 7 Tbili results, and change in Tbili from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 17 | 10
mg/dL
  Screening | 1.2 (0.7) | 1.2 (0.8) | 1.5 (1.7)
  Day 7: number analyzed (Participants) | 10 | 13 | 9
  Day 7 | 0.6 (0.2) | 0.6 (0.3) | 1.1 (0.8)
  Change from Screening to Day 7: number analyzed (Participants) | 10 | 13 | 9
  Change from Screening to Day 7 | -0.8 (0.6) | -0.5 (0.5) | -0.4 (1.4)

7. Primary Outcome: Serum Creatinine (sCr)
Description: Screening sCr results, Day 7 sCr results, and change in sCr from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 17 | 11
mg/dL
  Screening | 1.2 (0.5) | 1.2 (1.0) | 1.2 (0.7)
  Day 7: number analyzed (Participants) | 13 | 15 | 10
  Day 7 | 1.1 (0.9) | 1.3 (1.7) | 1.0 (0.4)
  Change from Screening to Day 7: number analyzed (Participants) | 13 | 15 | 10
  Change from Screening to Day 7 | -0.1 (0.7) | 0.1 (2.0) | -0.2 (0.6)

8. Primary Outcome: Albumin (Alb)
Description: Screening Alb results, Day 7 Alb results, and change in Alb from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 12 | 15 | 9
g/dL
  Screening | 2.5 (0.9) | 2.1 (0.5) | 2.3 (0.5)
  Day 7: number analyzed (Participants) | 10 | 12 | 8
  Day 7 | 1.9 (0.9) | 1.7 (0.4) | 2.3 (0.6)
  Change from Screening to Day 7: number analyzed (Participants) | 10 | 12 | 8
  Change from Screening to Day 7 | -0.6 (0.4) | -0.3 (0.2) | 0.1 (0.7)

9. Primary Outcome: Hemoglobin (Hgb)
Description: Screening Hgb results, Day 7 Hgb results, and change in Hgb from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 17 | 11
g/dL
  Screening | 11.5 (2.2) | 11.0 (1.5) | 10.5 (2.6)
  Day 7: number analyzed (Participants) | 13 | 14 | 10
  Day 7 | 8.8 (2.1) | 8.9 (1.1) | 9.0 (1.4)
  Change from Screening to Day 7: number analyzed (Participants) | 13 | 14 | 10
  Change from Screening to Day 7 | -2.9 (2.1) | -2.5 (1.5) | -1.3 (2.4)

10. Primary Outcome: Total White Blood Cell (WBC) Count
Description: Screening WBC results, Day 7 WBC results, and change in WBC from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: thousand cells per microliter
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 17 | 11
thousand cells per microliter
  Screening | 17.8 (10.0) | 14.7 (8.8) | 21.7 (16.2)
  Day 7: number analyzed (Participants) | 13 | 14 | 10
  Day 7 | 14.3 (6.7) | 12.5 (5.1) | 12.3 (2.4)
  Change from Screening to Day 7: number analyzed (Participants) | 13 | 14 | 10
  Change from Screening to Day 7 | -5.0 (9.3) | -3.0 (10.9) | -11.2 (14.9)

11. Primary Outcome: Platelet (PLT) Count
Description: Screening PLT results, Day 7 PLT results, and change in PLT from screening to Day 7
Time Frame: Screening and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: thousand cells per microliter
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 17 | 11
thousand cells per microliter
  Screening | 300.2 (182.2) | 215.1 (82.0) | 255.3 (130.0)
  Day 7: number analyzed (Participants) | 13 | 15 | 10
  Day 7 | 401.5 (168.8) | 341.8 (140.6) | 318.3 (148.2)
  Change from Screening to Day 7: number analyzed (Participants) | 13 | 15 | 10
  Change from Screening to Day 7 | 81.8 (237.1) | 125.1 (144.6) | 49.9 (160.2)

12. Primary Outcome: International Normalized Ratio (INR)
Description: Screening INR results, Day 7 INR results, and change in INR from screening to Day 7. In general, the higher the INR value, the longer it takes for blood to form a clot.
Time Frame: Screening and Day 7
Population: The safety analysis population consisted of all randomized patients who received study drug. One of the 0.25 mg/kg patients did not have a Screening INR result. Participant numbers in some rows differ from the overall number analyzed due to missing data as conveyed in the number of participants in each treatment group within a row.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 17 | 11
unitless
  Screening | 1.29 (0.22) | 1.43 (0.33) | 1.41 (0.38)
  Day 7: number analyzed (Participants) | 11 | 12 | 9
  Day 7 | 1.2 (0.1) | 1.2 (0.1) | 1.3 (0.3)
  Change from Screening to Day 7: number analyzed (Participants) | 11 | 12 | 9
  Change from Screening to Day 7 | -0.1 (0.2) | -0.2 (0.3) | -0.2 (0.3)

13. Primary Outcome: QT Interval With Fridericia's Correction (QTcF)
Description: Pre-dose QTcF, post-dose QTcF, change in QTcF from pre-dose to post-dose
Time Frame: Pre-dose and up to 24 hours post-dose
Population: Safety population: all randomized patients who received study drug. The number of patients analyzed is the number of patients with non-missing data as noted in results.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 16 | 11
msec
  Pre-dose QTcF | 419.1 (39.3) | 401.8 (16.8) | 405.1 (38.6)
  Post-dose QTcF: number analyzed (Participants) | 15 | 16 | 10
  Post-dose QTcF | 409.2 (23.1) | 403.1 (39.3) | 407.4 (29.6)
  Change in QTcF from pre-dose to post-dose: number analyzed (Participants) | 15 | 16 | 10
  Change in QTcF from pre-dose to post-dose | -9.9 (37.2) | 1.3 (36.1) | 8.9 (31.0)

14. Primary Outcome: Categorical Change in QTcF
Description: Number and percentage of patients with a change in QTcF of > 30 msec; number and percentage of patients with a change in QTcF of > 60 msec
Time Frame: Pre-dose and up to 24 hours post-dose
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 16 | 10
Participants
  Patients with a change in QTcF of > 30 msec | 1 | 3 | 2
  Patients with a change in QTcF of > 60 msec | 1 | 2 | 1

15. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Area under the plasma concentration versus time curve (AUC) from time zero to infinity following a single dose of study drug, obtained by noncompartmental methods. It is an integrated measure of study drug plasma exposure.
Time Frame: Prior to infusion, at mid infusion time, end of infusion, and at 2, 5, 10, 20, 30, 60 min and 120 minutes after completion of the IV infusion of study drug.
Population: The pharmacokinetic (PK) analysis population consisted of all intent-to-treat (ITT) patients who received study drug and had a baseline and at least one post-baseline specified plasma sample obtained for quantitative analysis. The number of subjects analyzed reflects the number of subjects for which the parameter could be determined.
Measure: Median (Full Range); unit: ng*min/mL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg
Number analyzed (Participants) | 7 | 14
ng*min/mL | 8497 [2836 to 14269] | 16921 [4843 to 28952]

16. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration (observed)
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: ng/mL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg
Number analyzed (Participants) | 11 | 16
ng/mL | 899 [98 to 2664] | 1484 [661 to 3418]

17. Primary Outcome: Apparent Terminal Plasma Half-life (T1/2)
Description: Apparent terminal plasma half-life (T1/2) is the amount of time for plasma concentrations to decline by 50%.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: minutes
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg
Number analyzed (Participants) | 7 | 14
minutes | 2.61 [1.28 to 18.99] | 4.89 [1.53 to 14.16]

18. Primary Outcome: Clearance (CL)
Description: Clearance (CL) is the volume of plasma completely cleared of drug per unit of time.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: mL/min/kg
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg
Number analyzed (Participants) | 7 | 14
mL/min/kg | 29.42 [17.52 to 88.14] | 29.55 [17.27 to 103.24]

19. Primary Outcome: Apparent Volume of Distribution Under Steady State Conditions (Vss)
Description: Apparent volume of distribution under steady state conditions (Vss) based on drug concentration in plasma
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: mL/kg
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg
Number analyzed (Participants) | 7 | 14
mL/kg | 100 [53 to 157] | 135 [36 to 318]

20. Secondary Outcome: C-reactive Protein (CRP)
Description: Screening CRP results, Day 7 CRP results, and change in CRP from screening to Day 7
Time Frame: Screening and Day 7
Population: The population is all randomized patients who received study drug. The number of patients analyzed is the number of patients with non-missing data in this population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 16 | 11
mg/dL
  Screening | 29.2 (12.3) | 27.5 (6.2) | 20.6 (13.2)
  Day 7 | 11.7 (10.0) | 7.5 (4.4) | 4.0 (3.0)
  Change from Screening to Day 7 | -19.2 (14.6) | -22.7 (5.9) | -20.5 (11.0)

21. Secondary Outcome: Day 14 Sequential Organ Failure Assessment (SOFA) Score
Description: Day 14 SOFA score is the sum of individual SOFA score components at Day 14. Results include last observation carried forward (LOCF) imputation for missing values.
  SOFA total scores range from 0 to 24, with higher scores reflecting a worse clinical status or outcome. A SOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
Time Frame: 14 days
Population: Modified intent-to-treat (mITT) population: all randomized patients who received the proper study drug (AB103 or Placebo), had a definitive surgical diagnosis of NSTI, were not mis-dosed, and did not have a CD4 count <200 cells/mm3. Proper study drug administration meant that study drug administration did not deviate from the planned administration.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 14 | 10
score on a scale | 1.07 (1.00) | 0.71 (0.83) | 2.70 (2.79)
Statistical Analysis 1: Comparison: AB103 0.25 mg/kg vs AB103 0.5 mg/kg vs Placebo; Test type: Other; p = 0.016, ANOVA

22. Secondary Outcome: Day 14 Sequential Organ Failure Assessment (SOFA) Score Less Than or Equal to 1
Description: Number and percentage of patients with Day 14 Sequential Organ Failure Assessment (SOFA) score less than or equal to 1. SOFA total scores range from 0 to 24, with higher scores reflecting a worse clinical status or outcome. A SOFA total score of 0 or 1 reflects resolution of organ dysfunction/failure.
Time Frame: 14 days
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 14 | 14 | 10
Participants | 10 | 13 | 4
Statistical Analysis 1: Comparison: AB103 0.25 mg/kg vs AB103 0.5 mg/kg vs Placebo; The null hypothesis was that the frequency of Day 14 SOFA score less than or equal to 1 was not different among treatment groups; Test type: Other; p = 0.019, Chi-squared

23. Secondary Outcome: Hospital Length of Stay (LOS)
Description: The duration of hospital stay over the 28-day study period.
Time Frame: 28 days
Population: Modified intent-to-treat (mITT) population: all randomized patients who received the proper study drug (AB103 or Placebo), had a definitive surgical diagnosis of NSTI, were not mis-dosed, and did not have a CD4 count <200 cells/mm3. Proper study drug administration meant that study drug administration did not deviate from the planned administration. The number of patients analyzed is the number of patients with non-missing data in this population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 10
days | 17.1 (7.96) | 17.4 (9.07) | 20.0 (6.93)
Statistical Analysis 1: Comparison: AB103 0.25 mg/kg vs AB103 0.5 mg/kg vs Placebo; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney) — Wilcoxon p value represents comparison of active dose groups versus placebo group

24. Secondary Outcome: Intensive Care Unit-free Days (ICU-free Days)
Description: The number of intensive care unit-free days (ICU-free days)
Time Frame: 28 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ICU-free days
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 10
ICU-free days | 21.7 (8.48) | 21.3 (6.21) | 17.1 (9.88)
Statistical Analysis 1: Comparison: AB103 0.25 mg/kg vs AB103 0.5 mg/kg vs Placebo; Test type: Other; p = 0.18, Wilcoxon (Mann-Whitney) — Wilcoxon p value represents comparison of active dose groups versus placebo group

25. Secondary Outcome: Ventilator-free Days
Description: The number of ventilator-free days (days without ventilator use)
Time Frame: 28 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ventilator-free days
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 10
ventilator-free days | 23.5 (8.75) | 24.1 (6.25) | 20.8 (9.14)
Statistical Analysis 1: Comparison: AB103 0.25 mg/kg vs AB103 0.5 mg/kg vs Placebo; Test type: Other; p = 0.19, Wilcoxon (Mann-Whitney) — Wilcoxon p value represents comparison of active dose groups versus placebo group

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) included in this summary were to be collected from dosing through Day 7; serious adverse events (SAEs) included in this summary were to be collected from dosing through Day 28.
Description: General, non-directed, systematic questioning of patients regarding AEs was to be performed at each study visit through Day 7. After Day 7, SAEs were to be assessed at each study visit through Day 28. Patients were able to voluntarily report AEs at any time.
Arm/Group | AB103 0.25 mg/kg | AB103 0.5 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/17 | 2/11
Serious Adverse Events (participants affected / at risk) | 8/15 | 5/17 | 4/11
Other Adverse Events (participants affected / at risk) | 14/15 | 16/17 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB103 0.25 mg/kg (N=15) | AB103 0.5 mg/kg (N=17) | Placebo (N=11)
Hypotension (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 1 (1) | 0 (0)
Withdrawal of life support (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Operative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Finger amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fungemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AB103 0.25 mg/kg (N=15) | AB103 0.5 mg/kg (N=17) | Placebo (N=11)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Face edema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Generalized edema (General disorders) | 0 | 0 | 1
Localized edema (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0
Edema peripheral (General disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 3 | 7 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Fungemia (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Operative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood (Investigations) | 0 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 5 | 6 | 3
Blood phosphorus decreased (Investigations) | 6 | 7 | 1
Blood potassium decreased (Investigations) | 5 | 7 | 3
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0
Clostridium test positive (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 0
Hematocrit decreased (Investigations) | 5 | 3 | 3
Haptoglobin increased (Investigations) | 1 | 0 | 0
International normalized ratio abnormal (Investigations) | 0 | 0 | 1
International normalized ratio increased (Investigations) | 0 | 0 | 1
Urine output decreased (Investigations) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 2
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Finger amputation (Surgical and medical procedures) | 1 | 0 | 0
Withdrawal of life support (Surgical and medical procedures) | 0 | 1 | 0
Arterial hemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 3 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No